CLINICAL TRIAL: NCT05071950
Title: The Effect of D-allulose on the Glycemic Changes in Patients With Type 2 Diabetes Mellitus During Ramadan Fasting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Collaborators: Matsutani Chemical Industry Co., Ltd. (Unknown); Kagawa University (Other)
Responsible Party: Principal Investigator, Salimah Binti Japar, RN, MPhil, Universiti Putra Malaysia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NMRR-19-3457-51288
Record Dates: First submitted 2021-09-27; First posted 2021-10-08 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Glucose, High Blood
Keywords: D-allulose; Ramadan fasting; Postprandial glucose; Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 14 days continuous glucose monitoring (Other): The participants started and completed the control period for continuous 7 days and followed with D-allulose period for 7 days
  Interventions: Other: Control period; Dietary Supplement: D-allulose period

INTERVENTIONS:
Other: Control period — * first 7 days, participants consumed normal meal during iftar (breaking the fast at sunset)
  * participants did not allow to have added sugar/ sweetness drinks before the iftar meal
  * flash continuous glucose monitoring system (FreeStyle Libre Pro) was used to measure the glucose
  * food diary was used to record the iftar meal
Dietary Supplement: D-allulose period — * [started after 7 days of control period],
  * participants continued with D-allulose period for 7 days continuously
  * participants consumed 8.5 g of D-allulose, (dissolve in plain water normal) before start the iftar meal
  * participants did not allow to have added sugar/ sweetness drinks before the iftar meal
  * flash continuous glucose monitoring system (FreeStyle Libre Pro) was used to measure the glucose
  * food diary was used to record the iftar meal
  * a questionnaire (multiple choice anwers) was used to record the side effects of D-allulose

SUMMARY:
Postprandial hyperglycemia or rapid rise in blood glucose is defined as a blood glucose level>7.8 mmol/L (140 mg/dL) 1- 2 hours after consumption of food. It is associated to the development of diabetes among healthy individuals and a risk factor for the onset and progression of microvascular and macrovascular complications among diabetic patients. In Ramadan, postprandial hyperglycemia is often observed after the iftar (fasting break after sunset). The frequency of eating normally decreases during Ramadan, however, the energy intake remains questionable because dietary practices during Ramadan are influenced by local culture, economic status and individual dietary behaviors. In many Muslim societies including Malaysia, Ramadan has known as a month of feasting. Iftar meals are typically high calorie, carbohydrate-rich and usually sweet food resulting in rapid rise in glucose after the meal. This poses a challenge for the people with diabetes to manage their glucose level. D-allulose (a C-3 epimer of D-fructose) is a rare sugar and reported to have several health benefits, such as suppressing a rise in postprandial glucose levels. There is still a scarcity of research on patients with diabetes. As a result, the current clinical study sought to investigate the effect of supplemental D-allulose on participants with type 2 diabetes who consume real-meal calories during Ramadan iftar.

DETAILED DESCRIPTION:
D-allulose (a C-3 epimer of D-fructose) is one of the rare sugar types with zero calories, has 70 % sweetness as sucrose, and occur in a small quantities in nature. Extensive basic and clinical studies have reported beneficial outcomes to human health, includes improve hypoglycemia, reduced postprandial hyperglycemia, hypolipidemia, and antioxidant. D-allulose can be taken up to 0.5 g/kg daily will no side-effect on the human body. The U.S. Food and Drug Administration (FDA) has declared that D-allulose is Generally Recognized As Safe (GRAS) for use as a food ingredient and with other sweeteners. Previous clinical studies on D-allulose had shown an effective glucose suppressive effect after the meal, mostly in healthy individuals and pre-diabetics. There is still a scarcity of research on patients with diabetes. As a result, the current clinical study sought to investigate the effect of supplemental D-allulose on participants with type 2 diabetes who consume real-meal calories during Ramadan iftar (breaking fast at sunset). This was a non-randomized intervention study, which involved a single-arm group, and conducted during Muslim fasting month (Ramadan) between 13 April to 12 May 2021. The protocol required continuous 14 days of Ramadan and it was divided into two consecutive periods; began with first 7-day of control period and followed with a consecutive 7-day of D-allulose period. At the D-allulose period, 8.5g of D-allulose was consumed before the iftar meal. The FreeStyle Libre Pro Flash Glucose Monitory system (CFGM) was used to measure the glucose values.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes (Group 4 -low-risk group as defined by International Diabetes Federation ) - low-risk group is defined as a well-controlled diabetic patient treated with lifestyle modification and oral anti-diabetic medications
* The patient was diagnosed with type 2 diabetes before the previous Ramadan. They also had fasted during previous year of Ramadan (2020) and are planning to fast during the coming Ramadan (2021)

Exclusion Criteria:

* Patients with poor glycemic control; HbA1c of 8% or more
* Patients with other serious complications
* Pregnant, maternal, breastfeeding or pregnant women
* Patients with severe renal dysfunction (serum creatinine level of 1.5 mg/dl or higher)
* Patients who advised not to fast by doctor
* Patients participating in other clinical trials
* Patients with contraindications to D-allulose

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Postprandial glucose (mg/dl) | 180 minutes
  * Evaluation on the effect of D-allulose on peak of postprandial glucose
  * the glucose levels were measured by flash continuous glucose monitoring system

SECONDARY OUTCOMES:
% TIR | 180 minutes
  Percentage of time glucose in-target range generated by flash continuous glucose monitoring system
% TAR | 180 minutes
  Percentage of time glucose above-target range generated by flash continuous glucose monitoring system
% TBR | 180 minutes
  Percentage of time glucose below-target range generated by flash continuous glucose monitoring system
side-effects of D-allulose | 24 hours
  Evaluate the side effects of D-allulose using a questionnaire [multiple choice answers]

CONTACTS AND LOCATIONS:
Overall Officials: Salimah Japar, Principal Investigator — Universiti Putra Malaysia
Locations (1):
- Universiti Putra Malaysia, Serdang, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Japar S, Fukunaga K, Kobayashi T, Imachi H, Sato S, Saheki T, Ibata T, Yoshimura T, Soh KL, Ong SL, Muhamed Z, Murao K. A pilot study on the effect of D-allulose on postprandial glucose levels in patients with type 2 diabetes mellitus during Ramadan fasting. Diabetol Metab Syndr. 2022 Jun 21;14(1):86. doi: 10.1186/s13098-022-00856-3. PMID 35729673